CLINICAL TRIAL: NCT05312216
Title: A Study on the Efficiency and Safety of Durvalumab Plus Lenvatinib as First-line Treatment for Unresectable Hepatocellular Carcinoma: an Open, Single Arm, Phase II Clinical Trial
Brief Title: Durvalumab Plus Lenvatinib as First-line Treatment for Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCLEPL1
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Durvalumab; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab plus Lenvatinib (Experimental): Durvalumab is a human IgG1 κ monoclonal antibody that inhibits binding of PD-L1 to its receptors PD-1 and CD80.
  Lenvatinib is a multi- kinase inhibitor of VEGF receptors 1 to 3, FGF receptors 1 to 4, PDGFRa, RET, and KIT.
  Interventions: Drug: Durvalumab plus Lenvatinib

INTERVENTIONS:
Drug: Durvalumab plus Lenvatinib — Durvalumab: 1500mg, iv.drip, Q4w Lenvatinib: 8mg, QD (body weight < 60kg) or 12mg, QD (body weight ≥ 60kg)
  Number of cycle: until subjects withdrawing the informed consent OR progressive disease OR developing unacceptable toxicity events

SUMMARY:
This is a phase II, open-label study to evaluate the efficacy and safety of Durvalumab plus Lenvatinib as first-line treatment in patients with unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
This single-arm, open-label, prospective phase II clinical trial was designed to evaluate the efficacy and safety of Durvalumab plus Lenvatinib as first-line treatment in patients with unresectable hepatocellular carcinoma. The primary endpoint is the objective response rate (ORR) according to RECIST v1.1. Safety evaluation will be taken according to CTCAE v5.0. Disease control rate (DCR), duration of response (DOR), progression-free survival (PFS) and overall survival (OS) are secondary endpoints. Multi-omics analysis will be performed to identify potential biomarkers for treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects volunteer to participate in the study and sign the informed consent before enrollment.
* 18-80 years of age.
* ECOG score of 0-1.
* Primary liver cancer with a pathological diagnosis of hepatocellular carcinoma.
* Child-Pugh grade A (5-6 points).
* BCLC C stage or BCLC B stage not suitable/refused for locoreginal treatments.
* Tumor volume ≤ 50% of the total liver volume.
* Without prior systemic therapy and unwilling to receive standard systemic therapy or unsuitable for standard systemic therapy.
* At least one measurable lesion as defined by RECIST v1.1 criteria.
* Patients infected with hepatitis virus should receive antiviral therapy regularly.
* No history of drug allergy.
* Function of vital organs in accordance with the following requirements (no blood components, cell growth factors and other corrective therapeutic agents are allowed within 14 days prior to enrolment): Absolute neutrophil count ≥ 1.5 x 10^9/L; Platelets ≥ 80 x 10^9/L; Haemoglobin ≥ 90 g/L; Serum albumin ≥ 35 g/L; Thyrotropin (TSH) ≤ 1×ULN (if abnormal, FT3 and FT4 levels should be examined at the same time, if FT3 and FT4 levels are normal, enrollment is allowed); Serum bilirubin ≤ 1.5 x ULN (within 7 days prior to first dose); ALT and AST ≤ 5 x ULN (within 7 days prior to first dose); International normalised ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 x ULN; Serum creatinine ≤ 1.5 x ULN.
* Female patients who are non-surgically sterilised or of childbearing age are required to use contraception (e.g. IUD, pill or condom) during and for 3 months after the end of the treatment; female patients of childbearing age who are non-surgically sterilised must have a negative serum or urine HCG test within 72h prior to study entry; and must be non-lactating; male patients whose partners are women of childbearing age should be tested during the trial and for 3 months after the last dose. Male patients whose partners are women of childbearing age should use an effective method of contraception during the trial and for 3 months after the last dose.

Exclusion Criteria:

* Patients with any active autoimmune disease or history of autoimmune disease (e.g. the following but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, autoimmune hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, vitiligo. Patients with complete remission of asthma in childhood who do not require any intervention in adulthood may be included, but those require bronchodilators cannot be included.
* Patients who are on immunosuppressive drugs, or require systemic hormone therapy for immunosuppression purposes (doses >10 mg/day of prednisone or other isotonic hormones) and who continue to use them within 2 weeks prior to enrollment.
* Receiving systemic therapy previously or other anti-cancer treatments (e.g. radiofrequency ablation, interventional therapy, radiotherapy, etc.)
* Patients with a known history of central neural system metastases or hepatic encephalopathy.
* Patients with clinically symptomatic ascites requiring puncture or drainage or those who have received ascites drainage within the previous 3 months.
* Patients with hypertension that is not well controlled by antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg).
* Having clinical cardiac symptoms or disease not well controlled, such as (1) NYHA class 2 or higher heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention (5) QTc > 450 ms (men); QTc > 470 ms (women).
* With abnormal coagulation (INR > 2.0, PT > 16s), bleeding tendency or on thrombolytic or anticoagulant therapy. Prophylactic use of low-dose aspirin or low molecular heparin is allowed.
* Patients had clinically significant bleeding symptoms or a clear bleeding tendency within the 3 months prior to enrollment.
* Having arterial/venous thrombotic events within the 6 months prior to enrollment.
* With hereditary or acquired bleeding and thrombotic tendencies.
* With urine protein ≥ ++ and confirmed by 24-hour urine protein amount > 1.0 g.
* Patients with active infection, unexplained fever ≥ 38.5°C within 7 days prior to the first dose, or baseline white blood cell count > 15 x 10^9/L.
* Patient with a congenital or acquired immune deficiency (e.g. HIV infection).
* Patient with other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) within the previous 3 years or concurrently.
* Patients who have other factors that could affect the outcome of the study or force the termination of the study, such as alcoholism, substance abuse, other serious illnesses (including psychiatric illness) requiring comorbid treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up o one year
  The proportion of patients who had tumor response evaluated as CR or PR according to RECIST v1.1 during study.

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to one year
  The proportion of patients who had tumor response evaluated as CR or PR or SD according to RECIST v1.1 during study.
Duration of response (DOR) | up to one year
  The duration from the first assessment of CR or PR to the first assessment of PD or death of any cause.
Progression-free survival (PFS) | up to one year
  The duration from the date of initial treatment to the date of disease progression (defined by RECIST v1.1) or death due to any cause.
Overall survival (OS) | up to two years
  The duration from the date of initial treatment to the date of death due to any cause.
Adverse events (AEs) | up to two years
  Any adverse events (including type, frequency and severity ) related with treatment drugs according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, PhD, Study Chair — Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No